CLINICAL TRIAL: NCT02618031
Title: The Capillary Index Score Trial: Phase I
Brief Title: The Capillary Index Score Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Firas Al-Ali (Other)
Collaborators: Stryker Neurovascular (Industry); Rochester General Hospital (Other); University of Vermont Medical Center (Other); University of North Carolina, Chapel Hill (Other); NYU Langone Health (Other); WellStar Health System (Other)
Responsible Party: Sponsor-Investigator, Firas Al-Ali, Neurointerventionalist, Cleveland Clinic Akron General
Organization: Cleveland Clinic Akron General (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CIS Trial
Record Dates: First submitted 2015-11-26; First posted 2015-12-01 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Acute Stroke; Brain Ischemia; Ischemic Stroke
Keywords: capillary index score; acute ischemic stroke; collateral circulation; cerebral ischemia; diagnostic imaging
MeSH Terms: conditions — Stroke; Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of two groups based on the outcome of diagnostic evaluation. Treatment will be identical for the two groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants and investigators evaluating 90 day outcomes will be blinded to the group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Favorable CIS (Other): Patients with a favorable CIS (fCIS) will receive endovascular treatment (EVT) and medical treatment consistent with national guidelines.
  Interventions: Procedure: Endovascular Treatment (EVT)
- Poor CIS (Experimental): Patients with a poor CIS (pCIS) will receive endovascular treatment (EVT) and medical treatment consistent with national guidelines.
  Interventions: Procedure: Endovascular Treatment (EVT)

INTERVENTIONS:
Procedure: Endovascular Treatment (EVT) — EVT is an endovascular procedure in which a catheter is inserted into an artery and directed to the site of the blocked blood vessel in the brain. The clot is removed using a mechanical device with or without an injection of tPA (tissue plasminogen activator) directly at the site of the clot. The protocol calls for use of the Trevo stent retriever (Stryker Neurovascular) for the first pass of clot removal.
  Other Names: Intra-arterial Treatment (IAT)

SUMMARY:
This study seeks to investigate the capillary index score (CIS) to further improve patient selection of endovascular treatment (EVT) in acute ischemic stroke (AIS).

The hypothesis or idea being tested:

Patients with favorable CIS who are successfully revascularized with EVT can have successful outcomes with an extended time window for treatment.

DETAILED DESCRIPTION:
This study is trying to look at how the well-being of the patient following treatment is influenced by peripheral blood supply (collateral flow) to the area lacking primary blood flow due to the clot. Treatment of AIS includes EVT and medical treatment. EVT is typically not offered to patients after 6 hours of the onset of symptoms. The current study is based on the belief that patients can be successfully treated with the EVT up to 8 hours, as long as they have good peripheral blood flow (collateral flow) to the area of tissue blocked of the primary blood supply.

The study will evaluate the ability of the capillar index score (CIS) to identify patients who can be successfully treated with EVT. The CIS quantifies blood supply to the ischemic area from peripheral vessels (collateral flow) based on diagnostic cerebral angiogram. Patients are graded on a scale from 0-3, with 0 and 1 considered a poor CIS (pCIS) and 2 and 3 considered a favorable CIS (fCIS). All patients will be treated with EVT and medical treatment consistent with national guidelines.

The primary endpoint is the clinical outcome at 90 days between fCIS group versus pCIS group. The secondary endpoint is the influence of successful revascularization on outcomes for patients with fCIS or pCIS.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior circulation acute ischemic stroke due to blockage of the intracranial internal carotid artery or middle cerebral artery (M1)
2. Within 24 hours of onset of symptoms
3. NIHSS Score is 8 or greater

Exclusion Criteria:

1. Contra-indication for IAT found on initial CT
2. Intracranial hemorrhage
3. Stroke mimics (tumor, herpetic encephalitis, etc.)
4. More than 1/3 hypodensity on non-enhanced head CT prior to intervention
5. ASPECT Score less than 6
6. Pre-existing disability defined as modified Rankin Scale (mRS) score more than 2
7. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Firas Al-Ali, MD, Principal Investigator — Cleveland Clinic Akron General
Locations (6):
- United States (6):
  - WellStar Atlanta Medical System, Atlanta, Georgia
  - New York University Langone Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- [Background] Al-Ali F, Elias JJ, Filipkowski DE, Faber JE. Acute ischemic stroke treatment, part 1: patient selection "the 50% barrier and the capillary index score". Front Neurol. 2015 Apr 22;6:83. doi: 10.3389/fneur.2015.00083. eCollection 2015. PMID 25954243
- [Background] Al-Ali F, Elias JJ, Filipkowski DE. Acute Ischemic Stroke Treatment, Part 2: Treatment "Roles of Capillary Index Score, Revascularization and Time". Front Neurol. 2015 Jun 1;6:117. doi: 10.3389/fneur.2015.00117. eCollection 2015. PMID 26082751
- [Background] Al-Ali F, Elias JJ, Tomsick TA, Liebeskind DS, Broderick JP; IMS Study Groups. Relative Influence of Capillary Index Score, Revascularization, and Time on Stroke Outcomes From the Interventional Management of Stroke III Trial. Stroke. 2015 Jun;46(6):1590-4. doi: 10.1161/STROKEAHA.115.009066. Epub 2015 May 7. PMID 25953374
- [Background] Al-Ali F, Tomsick TA, Connors JJ 3rd, Gebel JM, Elias JJ, Markarian GZ, Al-Ali Z, Broderick JP. Capillary Index Score in the Interventional Management of Stroke trials I and II. Stroke. 2014 Jul;45(7):1999-2003. doi: 10.1161/STROKEAHA.114.005304. Epub 2014 May 22. PMID 24851874
- [Background] Al-Ali F, Jefferson A, Barrow T, Cree T, Louis S, Luke K, Major K, Nemeth D, Smoker S, Walker S. The capillary index score: rethinking the acute ischemic stroke treatment algorithm. Results from the Borgess Medical Center Acute Ischemic Stroke Registry. J Neurointerv Surg. 2013 Mar;5(2):139-43. doi: 10.1136/neurintsurg-2011-010146. Epub 2012 Jan 19. PMID 22266703

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Final assignment to a group was not determined until the diagnostic cerebral angiograms were evaluated by the core lab at the end of the study to quantify the Capillary Index Score for each subject. Preliminary assessment of group was determined by the operators at the time of treatment.
Groups:
- Favorable CIS: Patients with a favorable CIS (fCIS) will receive endovascular treatment (EVT) and medical treatment consistent with national guidelines.
  Endovascular Treatment (EVT): EVT is an endovascular procedure in which a catheter is inserted into an artery and directed to the site of the blocked blood vessel in the brain. The clot is removed using a mechanical device with or without an injection of tPA directly at the site of the clot.
- Poor CIS: Patients with a poor CIS (pCIS) will receive endovascular treatment (EVT) and medical treatment consistent with national guidelines.
  Endovascular Treatment (EVT): EVT is an endovascular procedure in which a catheter is inserted into an artery and directed to the site of the blocked blood vessel in the brain. The clot is removed using a mechanical device with or without an injection of tPA directly at the site of the clot.
Period: Overall Study
Arm/Group | Favorable CIS | Poor CIS
Started | 46 | 11
Completed | 45 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: The core lab was unable to evaluate the CIS from the saved diagnostic cerebral angiograms for some of the enrolled subjects.
Groups:
- Favorable CIS: Patients with a favorable Capillary Index Score (fCIS) will receive endovascular treatment (EVT) and medical treatment consistent with national guidelines.
  Endovascular Treatment (EVT): EVT is an endovascular procedure in which a catheter is inserted into an artery and directed to the site of the blocked blood vessel in the brain. The clot is removed using a mechanical device with or without an injection of tissue plasminogen activator (tPA) directly at the site of the clot.
- Poor CIS: Patients with a poor Capillary Index Score (pCIS) will receive endovascular treatment (EVT) and medical treatment consistent with national guidelines.
  Endovascular Treatment (EVT): EVT is an endovascular procedure in which a catheter is inserted into an artery and directed to the site of the blocked blood vessel in the brain. The clot is removed using a mechanical device with or without an injection of tissue plasminogen activator (tPA) directly at the site of the clot.
- Total: Total of all reporting groups
Arm/Group | Favorable CIS | Poor CIS | Total
Number analyzed (Participants) | 46 | 11 | 57
Age, Continuous [Mean (Full Range); unit: years] | 70 [29 to 95] | 73 [44 to 86] | 70 [29 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 7 | 40
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 46 | 11 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 41 | 9 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 11 | 57
Height [Mean (Standard Deviation); unit: cm] | 165 (14) | 171 (6) | 166 (13)
Weight [Mean (Standard Deviation); unit: kg] | 82 (25) | 95 (20) | 85 (24)
diabetes [Count of Participants; unit: Participants] | 7 | 3 | 10
blood pressure [Mean (Standard Deviation); unit: mm Hg] | 147 (32) | 156 (32) | 149 (32)
occlusion site [Count of Participants; unit: Participants]
  middle cerebral artery (MCA) | 31 | 4 | 35
  internal carotid artery (ICA) | 2 | 1 | 3
  combination | 13 | 6 | 19
ischemic site [Count of Participants; unit: Participants]
  MCA | 41 | 6 | 47
  ICA | 1 | 1 | 2
  combination | 4 | 4 | 8
National Institutes of Health stroke scale [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health Stroke Scale provides a quantitative measure of stroke-related neurologic deficit. The scale includes 11 categories, graded on ability of the patient. The score ranges from 0 to 42, with 0 indicating normal function.
  units on a scale | 17 (5) | 21 (7) | 18 (6)

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Score (mRS) Between Favorable CIS Group Versus Poor CIS Group.
Description: The mRS Score ranges from 0-6 and describes the degree of disability or dependence after a stroke. The grades are no symptoms (0), no significant disability (1), slight disability (2), moderate disability (3), moderately severe disability (4), severe disability (5), and death (6).
Time Frame: 90 days
Population: A good outcome is defined as mRS 0-2
Measure: Count of Participants; unit: Participants
Arm/Group | Favorable CIS | Poor CIS
Number analyzed (Participants) | 45 | 11
Participants
  mRS 0-2 | 22 | 1
  mRS 3-6 | 23 | 10

2. Secondary Outcome: Complication Rate Between Favorable CIS Group Versus Poor CIS Group
Description: Complication : Clinically relevant intracranial hemorrhage and vasogenic edema as defined by parenchymal hematoma (PH) 1 or 2
Time Frame: 1 day - 1 week
Population: post-operative bleeding was not available for two subjects who died before a postoperative scan
Measure: Count of Participants; unit: Participants
Arm/Group | Favorable CIS | Poor CIS
Number analyzed (Participants) | 45 | 10
Participants
  PH 1 or 2 | 1 | 4
  no PH1 or 2 | 44 | 6

3. Secondary Outcome: Modified Rankin Score (mRS) Between Favorable CIS With Good Revascularization Versus Poor CIS With Good Revascularization.
Description: Revascularization status will be classified as poor (mTICI = 0-2A) or good (mTICI = 2B, 3). Rate of good clinical outcomes between groups will be compared based on the combination of CIS and revascularization status. Good outcome will be measured based on the modified Rankin scale score according to:
  0: No symptoms
  1. No significant disability despite symptoms
  2. Slight disability
  3. Moderate disability
  4. Moderately severe disability
  5. Severe disability
  6. Dead A score of 0-2 is considered a good outcome
Time Frame: 90 days
Population: output = number of patients with a good outcome one patient was lost to follow up
Measure: Count of Participants; unit: Participants
Groups:
- Favorable CIS and Good Revascularization: Patients with a favorable CIS (fCIS) who achieve good revascularization based on modified treatment in cerebral infarction (mTICI) score of 2B or 3
  Following endovascular treatment (EVT), revascularization was graded based on the mTICI classification according to:
  grade 0: no perfusion grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion grade 2A: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory grade 2B: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches
- Poor CIS and Good Revascularization: Patients with a poor CIS (pCIS) who achieve good revascularization based on modified treatment in cerebral infarction (mTICI) score of 2B or 3
  Following endovascular treatment (EVT), revascularization was graded based on the mTICI classification according to:
  grade 0: no perfusion grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion grade 2A: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory grade 2B: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches
- Favorable CIS and Poor Revascularization: Patients with a favorable CIS (fCIS) who achieve poor revascularization based on modified treatment in cerebral infarction (mTICI) score of 0, 1, or 2A
  Following endovascular treatment (EVT), revascularization was graded based on the mTICI classification according to:
  grade 0: no perfusion grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion grade 2A: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory grade 2B: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches
- Poor CIS and Poor Revascularization: Patients with a poor CIS (pCIS) who achieve poor revascularization based on modified treatment in cerebral infarction (mTICI) score of 0, 1, or 2A
  Following endovascular treatment (EVT), revascularization was graded based on the mTICI classification according to:
  grade 0: no perfusion grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion grade 2A: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory grade 2B: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches
Arm/Group | Favorable CIS and Good Revascularization | Poor CIS and Good Revascularization | Favorable CIS and Poor Revascularization | Poor CIS and Poor Revascularization
Number analyzed (Participants) | 36 | 8 | 9 | 3
Participants
  Good outcome | 19 | 1 | 3 | 0
  Poor outcome | 17 | 7 | 6 | 3

ADVERSE EVENTS:
Time Frame: 3 months
Description: All subjects in the study are considered at risk for death due to the nature of the stroke.
Arm/Group | Favorable CIS | Poor CIS
All-Cause Mortality (participants affected / at risk) | 8/45 | 7/11
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/11
Other Adverse Events (participants affected / at risk) | 2/45 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favorable CIS (N=45) | Poor CIS (N=11)
hemorrhage (Vascular disorders) | 1 (1) | 0 — Subarachnoid hemorrhage related to vessel perforation during treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Favorable CIS (N=45) | Poor CIS (N=11)
radiation (General disorders) | 2 (2) | 1 (1) — For three subjects at one site, the consent form did not adequately represent use of additional angiograms (100 milligrays of radiation) and contrast dye (20 mL) above standard of care for the site.

LIMITATIONS AND CAVEATS:
The sample size was limited by funding available to support the trial. The assignment of Capillary Index Score (CIS) by an independent core lab at the end of the trial led to a lower number of subjects in the poor CIS group than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02618031/Prot_SAP_000.pdf